CLINICAL TRIAL: NCT05888311
Title: Randomized, Open Clinical Study to Evaluate the Protective Potential of a Liquid Bandage Based on Liquid Elastic Collodion Versus no Treatment
Brief Title: Evaluation of the Protection of a Liquid Bandage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 184B
Record Dates: First submitted 2023-05-04; First posted 2023-06-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Skin Care
Keywords: effectiveness; Contact test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid bandage (Experimental): The liquid bandage will be applied after the tape strriping procedure and will be reapplied after 12 hours.
  Interventions: Device: Liquid bandage
- Control area (No Intervention)

INTERVENTIONS:
Device: Liquid bandage — Liquid elastic collodion- and benzethonium chloride-based topical solution
  Arms: Liquid bandage

SUMMARY:
This study was designed with the objective of evaluating the protection potential provided by the experimental product (Liquid Bandage) by evaluating its barrier formation capacity. Once the product's ability to form a barrier is confirmed, its ability to protect against small skin injuries, such as small cuts and bruises, blisters and cracks, is confirmed. The barrier formation also guarantees protection against the formation of calluses.

ELIGIBILITY:
Inclusion criteria

* Age between 18 and 70 years old.
* Fitzpatrick skin phototype classification I to IV.
* Presence of intact skin in the test region (right forearm and left forearm for selected participants).
* Agreement to adhere to the study procedures and requirements and attend the institute on the days and times determined for the assessments.
* Signing of the Informed Consent Form (ICF) and the Image Disclosure Consent Form (IDCF) before carrying out any study procedure.

Exclusion Criteria

* Diagnosis of skin diseases such as vitiligo, psoriasis, atopic dermatitis.
* Diagnosis of immunological insufficiency.
* Use of systemic corticosteroids or immunosuppressants.
* Diagnosis of type 1 diabetes mellitus or insulin-dependent diabetes or presence of complications resulting from diabetes (such as retinopathy, nephropathy, neuropathy), presence of diabetes-related dermatoses (such as plantar ulcers, lipoid necrobiosis, granuloma annulare, opportunistic infections), history of episodes of hypoglycemia, diabetic ketoacidosis and/or hyperosmolar coma.
* History of reaction to liquid dressings.
* Known hypersensitivity to any ingredients of investigational product formulation.
* Other diseases or use of drugs that may directly interfere with the study or put the research participant's health at risk.
* Presence of any serious or uncontrolled diseases, at the investigator's discretion.
* Pregnancy or lactation.
* Participation in a clinical research protocol in the last 12 months, unless, at the investigator's discretion, their participation in the study may result in direct benefit to the participant.
* Presence of any conditions that, at the investigator's discretion, make the participant unable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Efficacy of the investigational product in barrier formation, showing its superiority versus no treatment (control) through transepidermal water loss 12 hours after its administration. | 12 hours
  Evaluation of barrier formation through transepidermal water loss range 12 hours (± 20 minutes) after the end of tape stripping (TEWL12h) versus the measurement obtained immediately after tape stripping (TEWL0).

SECONDARY OUTCOMES:
Evaluate the efficacy of the investigational product in barrier formation through the range of transepidermal water loss 3 minutes after its administration | 3 minutes
  Evaluation of barrier formation through transepidermal water loss range 3 (±1) minutes after the end of tape stripping (TEWL3min) versus the measurement obtained immediately after tape stripping (TEWL0)
Evaluate the efficacy of the investigational product in barrier formation through the range of transepidermal water loss 6 hours after its administration. | 6 hours
  Evaluation of barrier formation through transepidermal water loss range 6 hours (± 10 minutes) after the end of tape stripping (TEWL6h) versus the measurement obtained immediately after tape stripping (TEWL0)
Evaluate the efficacy of the investigational product in barrier formation through the range of transepidermal water loss 24 hours after its administration | 24 hours
  Evaluation of barrier formation through transepidermal water loss range 24 hours (± 30 minutes) after the end of tape stripping (TEWL6h) versus the measurement obtained immediately after tape stripping (TEWL0)
Evaluate the efficacy of the investigational product in barrier formation through the range of corneometry 3 minutes after its administration | 3 minutes
  Evaluation of barrier formation through corneometry range 3 (± 1) minutes after the end of tape stripping (CM3min) versus the measurement obtained immediately after tape stripping (CM0)
Evaluate the efficacy of the investigational product in barrier formation through the range of corneometry 6 hours after its administration | 6 hours
  Evaluation of barrier formation through corneometry range 6 hours (± 10 minutes) after the end of tape stripping (CM6h) versus the measurement obtained immediately after tape stripping (CM0)
Evaluate the efficacy of the investigational product in barrier formation through the range of corneometry 12 hours after its administration | 12 hours
  Evaluation of barrier formation through corneometry range 12 hours (± 20 minutes) after the end of tape stripping (CM12h) versus the measurement obtained immediately after tape stripping (CM0)
Evaluate the efficacy of the investigational product in barrier formation through the range of corneometry 24 hours after its administration | 24 hours
  Evaluation of barrier formation through corneometry range 24 hours (± 30 minutes) after the end of tape stripping (CM24h) versus the measurement obtained immediately after tape stripping (CM0)
Evaluate the investigational product water resistance after four washes | 12 hours
  Water resistance as assessed by the average range of color change to activated charcoal pigment one (01), two (02), three (03), and four (04) washes after administration of the investigational product

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, Brazil